CLINICAL TRIAL: NCT03571139
Title: OCT Angiography Changes in Patients With Diabetes Mellitus Type 2 With and Without Diabetic Retinopathy Undergoing Phacoemulsification
Brief Title: Detecting the Influence of Cataract Surgery on the Development of Diabetic Retinopathy in Patients With Diabetes Mellitus Type 2 With and Without Diabetic Retinopathy Using OCT Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Tawfik Al Hanaineh, Doctor, Cairo University
Other Study IDs: Abeer T Al Hanaineh
Record Dates: First submitted 2018-06-15; First posted 2018-06-27 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Retinopathy
Keywords: OCT angiography; Diabetic retinopathy; Cataract surgery
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Diabetics type 2 with and without diabetic retinopathy: Patients with diabetes mellitus type 2 with and without diabetic retinopathy who needs cataract surgery by phacoemulsification. All patients will undergo OCT angiography examination prior to their cataract surgery and 4 weeks after the cataract surgery.
  Interventions: Device: Phacoemulsification

INTERVENTIONS:
Device: Phacoemulsification — Cataract surgery and in the bag posterior chamber lens implantation

SUMMARY:
Detecting the influence of cataract surgery on the development of diabetic retinopathy in patients with diabetes mellitus type 2 with and without diabetic retinopathy using OCT angiography.

DETAILED DESCRIPTION:
Patients with diabetes mellitus type 2 with and without without diabetic retinopathy (on biomicroscopy examination) who need cataract surgery, will undergo OCT angiography examination prior to their cataract surgery. Average vessel density (%) in superficial capillary plexus, deep capillary plexus and choriocapillaris, parafoveal vessel density (%) in the superficial and deep plexuses, FAZ area (mm2) in the superficial capillary plexus, FAZ circularity, retinal thickness, microaneurysms and capillary non-perfusion will be taken into analysis.

Patients will be examined on the first day after the cataract surgery with phacoemulsification and in the bag posterior chamber lens implantation.

All patients will undergo OCT angiography examination four weeks after their cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus type 2 with and without diabetic retinopathy who needs cataract surgery.
* Patients who need cataract surgery without any intravitreal injections.
* Absence of any ocular disease other than diabetes mellitus.
* Cataract density allowing good visualization of the fundus by OCT angiography.
* Patients with uneventful cataract surgery with phacoemulsification.

Exclusion Criteria:

* Patients who fail to comply with the follow-up schedule.
* Very dense cataract not allowing good visualization of the fundus by OCT angiography.
* Patients with complicated cataract surgery with phacoemulsification.
* Patients who need cataract surgery with any intravitreal injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus type 2 with and without diabetic retinopathy (on biomicroscopy examination) who need cataract surgery.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Detecting changes in the retinal vascular plexuses and choriocapillaris after cataract surgery in type 2 diabetes mellitus patients with and without diabetic retinopathy using OCT angiography. | 1 month
  Changes in the retinal vascular plexus, superficial and deep vessel density, foveal avascular zone area, circularity and any developing microaneurysms and areas of retinal ischemia will be measured to see the influence of cataract surgery on diabetic retinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer T Al Hanaineh, MSc, Principal Investigator — Cairo University
Locations (1):
- German Eye Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided